CLINICAL TRIAL: NCT00237874
Title: Aripiprazole Treatment of Prodromal Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YaleHIC26037
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Schizophrenia; Psychosis
Keywords: prodrome; ultra high risk; aripiprazole
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
We hypothesize that symptoms will improve in patients who meet diagnostic criteria for the schizophrenia prodrome when they are prescribed aripiprazole.

DETAILED DESCRIPTION:
This is an 8 week trial with extension for responders out to one year. All patients receive active medication; there is no placebo. Patients must meet criteria for the schizophrenia prodrome according to the Structured Interview for Prodromal Syndromes. Patients receive counseling as well. All counseling and medication are free of charge.

ELIGIBILITY:
Inclusion Criteria:

* age 13 to 40 meet criteria for the prodrome for schizophrenia

Exclusion Criteria:

* history of psychosis

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2004-02; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Total Score of the Scale Of Prodromal Symptoms | 8 weeks
  This is a 19-item scale with items scores 0-6. Treatment response is defined as all 5 Scale of Prodromal Syndromes positive symtpom items being rate below the prodromal range (< or equal to 2).

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Woods, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Institute of Living, Hartford, Connecticut
  - Yale School of Medicine, New Haven, Connecticut